CLINICAL TRIAL: NCT02669238
Title: Evaluation of a Subcutaneous Progestogen Implants in the Medical Management of Painful Endometriosis
Acronym: END-IMPACT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/CHU/03
Record Dates: First submitted 2015-10-22; First posted 2016-02-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant (Experimental): Subcutaneous insertion of an progestative implant containing 68mg of etonogestrel
  Interventions: Device: Nexplanon®
- Oral treatment (Active Comparator): Continuous oral administration of second generation monophasic oestro-progestative (ethinyl-oestradiol)
  Interventions: Drug: Minidril®/Leeloo®

INTERVENTIONS:
Device: Nexplanon® — Subcutaneous implant (Nexplanon®) containing etonogestrel 68 mg
  Arms: Implant
Drug: Minidril®/Leeloo® — continuous per os administration of oestroprogestative treatment. 1 pill a day First line: Minidril® (Levonogestrel 0.15 mg / Ethinylestradiol 0.03 mg) Second line: Leeloo® (Levonogestrel 0.1 mg / Ethinylestradiol 0.02 mg)
  Arms: Oral treatment

SUMMARY:
Endometriosis is a chronic relapsing disease characterized by the presence and proliferation of endometrial glands and stroma outside the uterus. This is a serious disease, widespread, difficult to live with for the patients, but also difficult to treat for practitioners who take care of these patients. It affects 1.6% of the general population, but its incidence is 10 times higher (up 40%) in patients with infertility. It occurs mainly by complex chronic pelvic pain and a negative influence on fertility.

It is a disease whose complexity can be explained to four levels. Firstly, through its extremely polymorphic character with intraperitoneal superficial forms, ovarian forms and deep sub-peritoneal forms.

Secondly by the plurality of the main symptoms which are individually non-specific and the frequency and / or intensity is not correlated with the severity of the disease. This non-specificity of symptoms partially explains the long lead misdiagnosis, which vary by 5 to 11 years.

Thirdly, by its prevalence which seems very high and largely underestimated. If its precise estimate in the general population is so complicated, it seems very high in many studies of patients supported surgically for gynecological reasons. These very large prevalence figures are observed when some consultations support the hypothesis of a widespread and probably insufficiently evaluated disease.

Lately by its management, insufficiently amended, for which there is currently only a few scientifically supported recommendations.

Chronic pain caused by the disease associated with altered sexuality to a loss of fertility significantly impacts the quality of life of patients.

DETAILED DESCRIPTION:
Investigators propose a randomized trial comparing two medical alternatives: a continuous monophasic type of estrogen-progestin oral treatment of second generation versus the establishment of an etonogestrel contraceptive implant type.

Are excluded from this study certain absolute surgical indications. Patients, by consenting to participate in the study, choose a medical care, which means not to be operated immediately. They are clearly informed about the various possible treatment alternatives. The benefits and risks of surgery and medical treatment they are explicitly presented. At any time during the study, patients who wish may discuss again a surgical treatment with their physician and stop the study drug if the decision of an intervention is taken.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years old
* with a painful symptomatic endometriosis
* with symptoms evolve for more than 6 months
* diagnosis based on clinical and radiological criteria : pain in the examination and/or palpation of endometriosis lesion(s) and lesion(s) objectified by MRI performed and interpreted by a radiologist referent dating less than three months at the time of inclusion
* no history presenting therapeutic surgery for endometriosis
* Accepting medical management
* without hormonal treatment (oestroprogestative, progestative or Luteinizing Hormone-Releasing Hormone (LHRH) analog) since at least 15 days
* No family history of deep venous thromboembolic disorders
* No abnormalities of hemostasis known
* Not pregnant at inclusion visit

Exclusion Criteria:

* Patient with a strict indication for surgery (ureteral disease with renal impact, digestive disease with occlusion, infertility with desire for immediate pregnancy, ovarian cyst ≥ 4cm)
* reproductive upper tract infections
* with one or more varicose veins
* with one or more breast abnormalities (ACR 3 or more)
* with contraindication for one of two treatments
* with contraindication for RMI
* taking drug treatment that could alter the concentration of the study treatments

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Global satisfaction | 6th month of treatment
  Global satisfaction evaluated by the SATMED-Q® satisfaction score at 6th month.

SECONDARY OUTCOMES:
Pain evaluation | 6th and 12th month
  Pain evaluation from analogical visual scale
Daily life impact | 6th and 12th month
  Evaluation of daily life impact of endometriosis with Endometriosis Health Profile - 30 (EHP-30)
Sex life impact | 6th and 12th month
  Evaluation of sexual life impact of endometriosis with Female Sexual Function Index (FSFI)
Evaluation of dysmenorrhea, dyspareunia and pelvic pain | 6th and 12th month
  Evaluation of frequency and intensity of dysmenorrhea, dyspareunia and pelvic pain with Biberoglu scale
Quality of life score | 6th and 12th month
  Evaluation of quality of life impact of endometriosis with SF36 scale
Number of lesions | Day 1 and 12th month
  The number, size, localisation and activity of the lesions is evaluated by Resonance Magnetic Image
size of lesions | Day 1 and 12th month
  Size of the lesions (mm) is evaluated by Resonance Magnetic Image
Localisation of lesions | Day 1 and 12th month
  Localisations of the lesions is evaluated by Resonance Magnetic Image
Incidence of treatment-emergent adverse events (safety and tolerability) | 3rd, 6th, 9th and 12th month
  percentage of clinical and biological adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Anca BIRSAN, MD, Principal Investigator
Locations (1):
- CHU de La Réunion, Saint-Denis, Saint Denis, Reunion

IPD SHARING:
Plan to Share IPD: No